CLINICAL TRIAL: NCT02165527
Title: Evaluation of Bone Length Measurement Using Lunar iDXA
Brief Title: Evaluation of Bone Length Measurement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Yebin Jiang, M.D., Principal Investigator, University of Michigan
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HUM29462
Record Dates: First submitted 2014-06-11; First posted 2014-06-17 (Estimated); Last update posted 2014-06-17 (Estimated); Status verified 2014-06

CONDITIONS: Bone Calcification; Osteoporosis
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- x-ray with iXDA scan (Experimental): Tota body scan taken by the Lunar iXDA. During the scan, subject will be asked to lay on their back. Following the Lunar iDXA scan, the computer of the Luna iXDA will calculate bone length. The calculation of bone length will be compared to a calculation from the subject's conventional x-ray to determine accuracy.
  Interventions: Procedure: Lunar iXDA scan

INTERVENTIONS:
Procedure: Lunar iXDA scan — Subject will receive a total body scan taken by the Lunar iXDA. This scan will take approximately 8 minutes to complete. Following the scan, the computer of the Lunar iXDA will calculate the bone length.

SUMMARY:
The purpose of this study is to determine if Lunar iXDA scanning with the use of a computer software program can make accurate measurements of the length of leg bones compared to conventional x-rays.

DETAILED DESCRIPTION:
The investigators would like to see how well the calculation of bone length using Lunar iDxa compares to conventional x-ray since the Lunar iXDA exposed patients to less radiation than conventional x-rays.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 yrs. of age or older
* Have recent x-rays of lower extremity
* Are at least 3 feet 7 inches tall and not taller than 6 feet 7 inches.

Exclusion Criteria:

* Are unwilling to read and sign the consent
* Are pregnant or if subject has not had a negative pregnancy test just prior to the iXDA scan
* Have severe deformities of your legs or back
* Unable to lay on the scanning table for the scan

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-11; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Leg (Femur and Tibia) bone length measurement in centimeters using iDXA | scan time is 8 minutes
  Lunar iXDA computer will calculate the bone length following a total body scan taken by the Lunar iDXA and compare results from conventional x-ray to determine accuracy.

CONTACTS AND LOCATIONS:
Overall Officials: Yebin Jiang, MD, PhD, Principal Investigator — University of Michigan Hospital
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States